CLINICAL TRIAL: NCT03408327
Title: The Application of Wearable Technology to Improve the Physical Activity Level of People With Chronic Mental Illness- Accuracy, Acceptability, Feasibility and Effectiveness Analysis
Brief Title: The Application of Wearable Technology to Improve the Physical Activity Level of People With Chronic Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-SV(I)-20150091
Record Dates: First submitted 2018-01-01; First posted 2018-01-24 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia; Physical Activity; Health Knowledge, Attitudes, Practice
Keywords: Schizophrenia; Physical Activity; Health Promotion; Wearable Technology; Fitness Wristband; mobile health, mHealth
MeSH Terms: conditions — Schizophrenia; Motor Activity; Behavior | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: We will conduct a single-blinded, randomized controlled study. Ninety participants will be randomly assigned to experimental group or control group. The intervention for both groups will last for 12 weeks, with a 12-week of follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Wearable technology (fitness wristband & App)
  2. 4 times group activities (2 hr / each times)
  3. LINE group interaction
  4. Reminder and feedback form researcher
  Interventions: Device: Wearable technology; Behavioral: LINE group; Behavioral: Group activities
- Control group (Active Comparator): 1. Wearable technology (fitness wristband + App)
  2. Health promotion manual
  Interventions: Device: Wearable technology; Device: Health promotion manual

INTERVENTIONS:
Device: Wearable technology — Fitness wristband & APP
Behavioral: LINE group — Promote social interaction
  Arms: Experimental group
Behavioral: Group activities — Which was developed by applying social cognitive theory
  Arms: Experimental group
Device: Health promotion manual — Which was about general physical activity promotion content
  Arms: Control group

SUMMARY:
The object is to develop a physical activity promotion program by applying social cognitive theory and wearable technology and evaluate its feasibility in people with MI

Stage I: Accuracy, Acceptability, Feasibility. Stage II: Effectiveness Analysis

In stage II, will conduct a single-blinded, randomized controlled study. 90 participants will be randomly assigned to experimental group or control group. The intervention for both groups will last for 12 weeks, with a 12-week of follow-up. The measurements include physical activity level, physical fitness, cognitive function and sleep quality, as well as the moderators of the effectiveness of program.

DETAILED DESCRIPTION:
Background: The health condition of individuals with chronic mental illness (MI) is usually poorer than the general population. This health disparity may be related to their lower physical activity level. One of the critical issues in psychiatric rehabilitation is to develop a health promotion program which utilizes less clinical resources and results in long-term effectiveness. Compared with structure exercise, lifestyle physical activity might be one of the solutions. With the mobile technology and wearable technology becoming popular, mobile health (mHealth) emerges and has showed some preliminary effects on other population. The mHealth may be an innovative health promotion program for people with MI and deserves more research to examine the effectiveness.

Purpose: This study is (1) to examine the accuracy and acceptability of wearable technology in persons with MI; (2) to develop a physical activity promotion program by applying social cognitive theory and wearable technology and evaluate its feasibility in people with MI ; (3) to examine the effectiveness of the program on physical activity level and health outcomes ; and (4) to examine the moderators of the program's effectiveness.

Methods:

Stage I: completed (Accuracy, Acceptability, Feasibility) Stage II: (RCT) The investigators will conduct a single-blinded, randomized controlled study. 90 participants will be randomly assigned to experimental group or control group. The intervention for both groups will last for 12 weeks, with a 12-week of follow-up. The measurements include physical activity level, physical fitness, cognitive function and sleep quality, as well as the moderators of the effectiveness of program.

Contributions: The results of study will be one of the evidence-based health promotion programs for individuals with MI. With wearable technology and telecommunication technology, it makes possible to expand the health care services from traditional clinical settings to client's natural milieu, and to serve more people with MI by using less resources. The results of study may also form a much appreciated basis for future studies of mHealth on other heath behavior (e.g., healthy diet) or in other disability groups (e.g., stroke).

ELIGIBILITY:
Inclusion Criteria:

1. having a diagnosis of SMI (including schizophrenia, depression, and bipolar disorder over one year) made by a psychiatrist on the basis of the criteria set Diagnostic and Statistical Manual of Mental Disorders, 5th edition, text-revision, DSM-V
2. living in the community and receiving community-based mental health rehabilitation services
3. having stable psychiatric conditions (i.e., primary psychiatric medications had not changed for more than two months)
4. being 20 to 64 years old
5. No obvious cognitive impairment (Mini-Mental Status Exam >24)
6. can follow the research process and sign the consent

Exclusion Criteria:

1. having a clinically significant physical condition making it unsafe to increase daily walking activity, such as severe coronary heart disease or musculoskeletal problems
2. according participants' self-statement, having following illness, including severe heart failure,myocardial infarction, angina pectoris, chronic obstructive pulmonary disease, COPD, poor glycemic control (i.e., dialysis, diabetic neuropathy or retinopathy) and lower extremity arthritis
3. uncontrolled hypertension with SBP> 160 mmHg or DBP> 110 mmHg
4. has significant cognitive impairment
5. unconscious or confused
6. already exercising regularly (i.e., doing moderate-intensity physical activities for 150 minutes each week)
7. participating in other intervention studies

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Objective daily physical activity data | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Using the fitness wristband App to view the daily step counts.

SECONDARY OUTCOMES:
Subjective daily physical activity data | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  International Physical Activity Questionnaire-Taiwan(IPAQ-TW), it is a self-reported questionnaire to survey participants' physical activity data in pass 7 days. There are total seven questions to check the physical activity time in seven life domains, including work, housework, gardening, transportation , leisure, exercise and siting activity. After the survey, researcher will convert the data in to quantitative data in order to calculate participants' metabolic equivalent (MET·min).
Body composition | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Using Body Mass Index (BMI) as the measurement of body composition, which weight and height will be combined to report BMI in kg/m^2.
Cardiorespiratory fitness | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Using 6-minute walk test (6MWT) as the measurement, which let the participant walk as far as possible over a total of six minutes on hard and flat floor. And researcher will measure the distance that participant walk in 6 minutes.
Muscular strength | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Hand-grip dynamometer to test the muscular strength of upper limb.The participant holds the dynamometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body. The units is in kg.
Leg muscular strength and endurance | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Using 30-Second Sit to Stand Test. The participant will sit in the middle of the chair, and rise to a full standing position, then sit back down again. Repeat this for 30 seconds.And researcher will count the times.
Balance and mobility | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  The Timed Up and Go test (TUG). It measure the time that the participant takes to rise from a chair, walk eight foots, turn around, walk back to the chair, and sit down.
Attention and processing speed | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Symbol digit modalities test (SDMT), which makes the participant to pair specific numbers with given geometric figures as fast as possible in 90 seconds. The researcher will record the total, correct and wrong answer numbers.
Verbal working memory | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Digit span test, which researcher will read a sequence of numerical digits, and the participant may to recall the sequence correctly. There are two part of this test, one is given forwards, other is backwards. these are in order to test the participant 's maximal memory span. Total scores is sum of forwards and backwards test, between 0 to 30.
Cognitive flexibility | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Stroop color word test. In this test, the participant will read out the color of the word as fast as possible. Instead of read the word meaning. The scoring is the number of correct answer.
Self-efficacy in exercise | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Self-Efficacy for Exercise Scale (SEES) is a self-report survey. It is used to evaluate the degree of participant's self-efficacy in exercise. There are total 9 descriptions, and participant will answer the degree of confidence (1-10 points). The scoring is used average as record, so the scale scores ranges is between 1 to 10. The higher values represent a better outcome.
Attitude to exercise | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Outcome Expectations for Exercise Scale (OEES) is a self-report survey. It is used to evaluate participant's attitude to exercise. There are total 9 descriptions, and participant will answer the degree of agreement. Statements are rated 1 (strongly disagree) to 5 (strongly agree). The total score is the sum of all nine items,so the scale scores ranges is between 9 to 45. The higher values represent a better outcome.
Behavior of exercise goal setting | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Exercise Goal Setting Scale (EGS) is a self-report survey. It is used to evaluate participant's attitude to exercise. There are total 10 descriptions, and participant will answer the degree of agreement. Statements are rated 1 (strongly disagree) to 5 (strongly agree). This scoring is used average as record, so the scale scores ranges is between 1 to 5. The higher values represent a better outcome.
The situation encountered during exercise | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Exercise Benefits/Barriers Scale (EBBS) is a self-report survey. It is used to evaluate 29 items of exercise benefits and 14 items of possible exercise barriers. There are total 43 descriptions, and participant will answer the degree of agreement. Statements are rated 1 (strongly disagree) to 4 (strongly agree). When the Benefits Scale is used alone, the score range is between 29 and 116.The higher the score, the more positively the individual perceives exercise. On the other hand, when the Barriers Scale is used alone, scores range between 14 and 56. If used alone, the higher the score on the Barriers Scale, the greater the perception of barriers to exercise.
The situation of social support | Change from baseline outcome measure at 12 weeks (post-test),and at 24 weeks (follow-up test)
  Social Support and Exercise Survey (SSES) is a self-report survey. It is used to evaluate participant's exercise performance change from family and friends' influence. There are 13 items of behaviors that family or friends do during last 3 months, which might be benefits or barriers of participant exercise regularly, and participant will answer the degree of frequency. Statements are rated 1 (none) to 4 (very often).The survey should be scored differently for friends and family. Family Participation: sum items 1~6 and 10~13 (scores ranges is between 10 to 40. The higher values represent a better outcome.)；Family Rewards and Punishment (an optional scale): sum items 7~9 (scores ranges is between 3 to 12. The lower values represent a better outcome.)；Friend Participation: sum items 1~6 and 10~13 (scores ranges is between 10 to 40. The higher values represent a better outcome.).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-De Chen, Ph.D., Principal Investigator — Department of Occupational Therapy, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No